CLINICAL TRIAL: NCT06520462
Title: Clinical Research of Comparative Effectiveness of Pharmacopuncture Therapy and Acupuncture Therapy for Chronic Neck Pain: A Pragmatic Randomized Strategy Comparative Clinical Trial
Brief Title: PCT of Pharmacopuncture for Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2024-01
Record Dates: First submitted 2024-07-22; First posted 2024-07-25 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Neck Pain; Chronic Pain
MeSH Terms: conditions — Neck Pain; Chronic Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacopuncture group (Experimental): 1. Acupoints: The selection of acupoints, depth of insertion, and other procedural details are determined based on the clinical judgment of the physicians according to the participant's symptoms, diagnostic imaging, and degree of improvement. Acupoints may include GB20, GB21, BL11, and EX-B2. However, these acupoints are not restrictive; any acupoints used for the treatment of chronic neck pain will be documented.
  2. Pharmacopuncture: The type and dosage of the pharmacopuncture solution used during treatment will be selected based on the clinical judgment of the physicians performing the pharmacopuncture. The types of pharmacopuncture solutions and the total amount administered will be recorded. The choice will be based on the participant's symptoms and the clinical judgment within the range of pharmacopuncture solutions currently used in clinical practice at the trial institution, without adding new solutions specifically for this study.
  Interventions: Procedure: Pharmacopuncture
- Acupuncture group (Active Comparator): The selection of acupoints, depth of insertion, and other procedural details are to be determined based on the clinical judgment of the physicians according to the participant's symptoms, diagnostic imaging, and degree of improvement. Acupoints may include sites such as GB21, SI9, GB20, GV14, and distal points like SI3. The number of needles used can range from 5 to 30. All acupoints treated during the procedure are to be documented.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Pharmacopuncture — The physicians will decide the specific methods of pharmacopuncture based on the clinical judgment according to each participant's conditions. All applied treatment methods are documented in the case report forms.
  Arms: Pharmacopuncture group
Procedure: Acupuncture — The physicians will decide the specific methods of acupuncture based on the clinical judgment according to each participant's conditions. All applied treatment methods are documented in the case report forms.
  Arms: Acupuncture group

SUMMARY:
A pragmatic clinical study to compare the effectiveness of pharmacopuncture and acupuncture treatment strategies in patients with chronic neck pain

DETAILED DESCRIPTION:
This study aims to confirm the comparative effectiveness of pharmacopuncture by conducting a pragmatic randomized controlled clinical trial with 128 patients suffering from chronic neck pain. The trial will compare patients treated with a pharmacopuncture-based strategy (64 patients) to those treated with an acupuncture-based strategy (64 patients). As this is a pragmatic clinical trial, participants will be randomly assigned to either the pharmacopuncture or acupuncture groups. However, the specific methods of pharmacopuncture and acupuncture to be used will not be predetermined. Instead, they will be determined based on the clinical judgment of the traditional Korean medicine doctor according to the patient's condition. All methods used will be recorded in the CRF (Case Report Form).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with neck pain persisting for more than 3 months
2. Patients with a Numeric Rating Scale (NRS) score of 5 or higher for neck pain
3. Patients aged between 19 and 70 years
4. Patients who agree to participate in the clinical study and provide a written informed consent form

Exclusion Criteria:

1. Patients diagnosed with serious specific diseases that could be the cause of neck pain (e.g., spinal metastasis of tumors, acute fractures, and spinal dislocations)
2. Patients exhibiting progressive neurological deficits or severe neurological symptoms
3. Patients whose pain originates from soft tissue disorders rather than the spine (e.g., tumors, fibromyalgia, rheumatoid arthritis, gout)
4. Patients with other chronic diseases that could interfere with the interpretation of treatment effects or outcomes (e.g., stroke, myocardial infarction, kidney disease, diabetic neuropathy, dementia, epilepsy)
5. Patients currently taking steroids, immunosuppressants, psychiatric medications, or other drugs that could affect the study results
6. Patients for whom pharmacopuncture treatment is inappropriate or unsafe: those with bleeding disorders, those undergoing anticoagulant therapy, and severe diabetic patients with infection risks
7. Patients who have taken medications that could affect pain (e.g., Non-Steroidal Anti-Inflammatory Drugs, NSAIDs) or received pharmacopuncture, acupuncture, or physical therapy within the past week
8. Pregnant women, those planning to become pregnant, or those currently breastfeeding
9. Patients who have undergone cervical spine surgery within the past 3 months
10. Patients who have not completed participation in another clinical study within the past month or plan to participate in another clinical study during the study participation and follow-up period within 6 months from the date of selection
11. Patients who find it difficult to provide informed consent for participation
12. Other cases where the researcher deems participation in the clinical study to be difficult

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Neck pain Numeric Rating Scale, NRS | Week 5
  Change from baseline to Week 5 on the Numeric Rating Scale of neck pain

SECONDARY OUTCOMES:
Neck and arm pain Numeric Rating Scale | Week 1,2,3,4,5,8,12
  The pain intensity of neck and arm over the past week
Neck and arm pain Visual Analogue Scale | Week 1,2,3,4,5
  The pain intensity of neck and arm over the past week
Northwick Park Questionnaire | Week 1,5,8,12
  A self-reported questionnaire consisting of 9 items related to the impact of neck pain on daily activities
Neck disability index | Week 1,5,8,12
  The degree of neck disability in daily life
Patient Global Impression of Change | Week 5,8,12
  The subject's subjective improvement
Health-related Quality of Life Instrument with 8 Items | Week 1,5,8,12
  A tool developed to measure the health-related quality of life in Koreans
5-Level EuroQol-5 Dimension | Week 1,5,8,12
  A tool that evaluates health status from multiple perspectives, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Adverse events | Week 1,2,3,4,5,8,12
  An undesirable and unintended sign, symptom, or disease that occurs after a procedure during the clinical study.

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, Study Director — Jaseng Medical Foundation
Locations (6):
- South Korea (6):
  - Daejeon Jaseng Hospital of Korean Medicine, Daejeon, Daejeon
  - Kyung Hee University Korean Medicine Hospital, Seoul, Dongdaemun-gu
  - Kyung Hee University Korean Medicine Hospital at Gangdong, Seoul, Gangdong-gu
  - Dongguk University Bundang Oriental Hospital, Seongnam, GGyeonggi-do
  - Bucheon Jaseng Hospital of Korean Medicine, Bucheon-si, Gyeonggi Province
  - Haeundae Jaseng Hospital of Korean Medicine, Busan

IPD SHARING:
Plan to Share IPD: No